CLINICAL TRIAL: NCT03161223
Title: Phase 1/2a Study of Anti-PD-L1 Monoclonal Antibody Durvalumab in Combination With Pralatrexate and Romidepsin, Oral 5-Aza and Romidepsin, Romidepsin Alone, or Oral 5-Azacitidine for Treatment of Patients With Relapsed and Refractory PTCL
Brief Title: Durvalumab in Different Combinations With Pralatrexate, Romidepsin and Oral 5-Azacitidine for Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAR0365
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma, T-Cell
Keywords: Durvalumab; Pralatrexate; Romidepsin; 5-Azacitidine
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — durvalumab; 10-propargyl-10-deazaaminopterin; romidepsin; Depsipeptides; Azacitidine

STUDY DESIGN:
Intervention Model Description: Phase 1 A minimum of 3 patients will be treated at the entry Dose Level, that is the MTD, in each arm. An estimated 10 patients will be accrued in each Arm, assuming ≤ 1 patients experience DLT. If a DLT is reached early we will treat fewer patients. For each study Arm, we will expand the MTD cohort to a total of 10 patients. We estimate that a total of 40 patients will be needed.
  Phase 2 Once the recommended phase 2 dose is identified, a planning meeting with the Sponsor and involved investigators will be convened to discuss which Arm(s) to advance to phase 2. The sample size of the phase 2 portion of the study will be calculated on an optimal 2-stage design. We will first enroll 8 patients. If at least 3 objective responses (PR or CR) are seen, then an additional 16 patients will be enrolled. If 10 or fewer patients respond, the combination will not be considered for further study. We will enroll a total of 24 patients per arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- A: Oral 5-azacitidine, durvalumab, romidepsin (Other): Arm A: Patients will first undergo a 7-day lead-in phase of 5-azacitidine. 5-azacitidine will be administered orally from day 1 to day 14 (including the lead-in phase), durvalumab will be administered intravenously on day 8 and romidepsin intravenously on days 8 and 15 of a 28-day treatment cycle
  Interventions: Drug: Durvalumab; Drug: Romidepsin; Drug: 5-Azacitidine
- B: durvalumab, pralatrexate, romidepsin (Other): Arm B: Durvalumab will be administered intravenously on day 1, pralatrexate will be administered intravenously on days 1 and 15, and romidepsin will be administered intravenously on days 1 and 15. Each treatment cycle will last 28 days. All patients receiving pralatrexate will receive folic acid and vitamin B12 supplementation according to the drug package insert. Leucovorin rescue is also allowed at the dose of 15 mg orally twice daily on days 3 to 6 and 17 to 20.
  Interventions: Drug: Durvalumab; Drug: Pralatrexate; Drug: Romidepsin
- C: durvalumab, romidepsin (Other): Arm C: Durvalumab will be administered intravenously on day 1 and romidepsin will be administered intravenously on days 1, 8, and 15 of a 28-day treatment cycle
  Interventions: Drug: Durvalumab; Drug: Romidepsin
- D: durvalumab, 5-azacitidine (Other): Arm D: Patients will first undergo a 7-day lead-in phase of 5-azacitidine. 5-azacitidine will be administered orally from day 1 to day 14 (including the lead-in phase) and durvalumab will be administered intravenously on day 8 of a 28-day treatment cycle
  Interventions: Drug: Durvalumab; Drug: 5-Azacitidine

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is an investigational human monoclonal antibody that works to inhibit (block) a protein called programmed cell death-1 ligand 1 (PD-L1). Durvalumab has not been approved by the FDA for the treatment of PTCL but has been given to patients other types of cancers. Given intravenously (through the vein).
  Starting dose: 1500 mg
  Other Names: MEDI4736
Drug: Pralatrexate — Pralatrexate is an antimetabolite drug. Pralatrexate alone is FDA-approved for the treatment of PTCL. Given intravenously (through the vein).
  Starting dose: 25 mg/m2
  Other Names: Folotyn
  Arms: B: durvalumab, pralatrexate, romidepsin
Drug: Romidepsin — Romidepsin is another type of chemotherapy known as histone deacetylase (HDAC) inhibitors. Romidepsin has not been approved for use in lymphoma other than Cutaneous T cell lymphoma (CTCL) by the FDA. Given intravenously (through the vein).
  Starting dose: 12 mg/m2
  Other Names: Depsipeptide
  Arms: A: Oral 5-azacitidine, durvalumab, romidepsin; B: durvalumab, pralatrexate, romidepsin; C: durvalumab, romidepsin
Drug: 5-Azacitidine — Oral 5-azacitidine is used for the treatment of myelodysplastic syndrome and acute myeloid leukemia. Azacitidine prevents the body from making DNA and RNA that cells need to grow. This stops the growth of cancer cells and causes them to die. Given by mouth (orally).
  Starting dose: 300 mg daily
  Other Names: Vidaza; Oral 5-Azacitidine
  Arms: A: Oral 5-azacitidine, durvalumab, romidepsin; D: durvalumab, 5-azacitidine

SUMMARY:
This is an open-label, Phase 1/2a, dose-finding study with an initial phase 1 portion, articulated in four separate treatment arms, followed by a dedicated phase 2 for qualifying treatment Arm(s).

The primary objective of the Phase 1 portion is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of: Durvalumab, oral 5-azacitidine, and romidepsin (Arm A); durvalumab, pralatrexate, and romidepsin (Arm B); durvalumab and romidepsin (Arm C); or durvalumab and oral 5-azacitidine (Arm D), in patients with peripheral T-cell lymphoma (PTCL). The safety and toxicity profile of these combinations will be evaluated throughout the entire study.

If one or more of the combinations in Arms A, B, C, or D are found to be feasible and an MTD is established, the phase 2 portion of the study will be initiated for the combination(s) with the strongest efficacy signal provided acceptable toxicity.

DETAILED DESCRIPTION:
The peripheral T-cell lymphomas (PTCL) are a heterogeneous group of aggressive lymphoid neoplasms and account for 10-15% of all newly diagnosed cases of non-Hodgkin's lymphoma (NHL). The current prevalence of PTCL in the United States is estimated to be approximately 9,500 patient. Treatment options for patients with relapsed/refractory (R/R) PTCL have been limited. This study focuses on exploring rational combinations of these T-cell active agents in an effort to develop novel treatment platforms.

ELIGIBILITY:
Inclusion Criteria (these criteria apply to both the phase 1 and phase 2 portion of the study)

* Age >18 years at the time of signing the informed consent
* Patients must have histologically confirmed newly diagnosed (ND) or Relapsed/Refractory Peripheral T-Cell Lymphoma (R/R PTCL) defined according to the 2016 World Health Organization (WHO) classification criteria.
* Patients with R/R PTCL who have received at least one previous line of therapy are eligible to be enrolled in this study.
* Patients who are candidate for an autologous or allogeneic stem cell transplantation (SCT) will be allowed to receive the study drugs as a "bridge" to transplantation.
* Evaluable (phase 1) or measurable (phase 2) disease.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients must have adequate organ and marrow function as defined by:

  1. Aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2 x institutional upper limit of normal (ULN); total bilirubin ≤ 1.5 x ULN (AST, ALT, and total bilirubin ≤ 3 × ULN in subjects with documented Gilbert's syndrome or hyperbilirubinemia clearly attributed to lymphoma involvement of the liver);
  2. Creatinine levels < 2 mg/dL; or creatinine clearance > 40 mL/min
  3. Absolute neutrophil count (ANC) > 1,000/μL; platelet count > 75,000/μL
  4. Negative urine or serum pregnancy test for women of childbearing potential. All women of childbearing potential must agree to use an effective barrier method of contraception (either an intrauterine device (IUD) or double barrier method using condoms or a diaphragm plus spermicide) during the treatment period and for at least 1 month after discontinuation of the study drugs. Male subjects should use effective barrier method of contraception during the treatment period and for at least 3 months after discontinuation of the study drugs.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria (these criteria apply to both the phase 1 and phase 2 portion of the study)

* Prior Therapy (for patients with R/R PTCL)

  1. Exposure to any agent targeting PD-1, PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4).
  2. For three-drug combinations, the patient must not have been exposed to at least two of those drugs. For two drugs combinations patients must not have been exposed to any of those drugs. Patients will be enrolled in the first treatment Arm that satisfies this exclusion criterion, according to the following sequence: Arm A; Arm B; Arm C; Arm D.
  3. Exposure to biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation therapy within 2 weeks prior to entering the study or lack of resolution of AE due to previously administered antineoplastic therapy to grade 1 or less according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.
  4. Current or prior use of immunosuppressive medication within 14 days prior to first dose of durvalumab. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10 mg/day of prednisone or equivalent for at least 5 days prior to the start of the study drugs.
  5. Prior allogeneic SCT
* History of, or suspected allergic reactions to, durvalumab, pralatrexate, oral 5-azacitidine, or romidepsin or any of their excipients.
* For patients who are treated with oral 5-azacitidine, any gastrointestinal disorder that would interfere with the absorption of the study drug
* Concomitant use of CYP3A4 inhibitors
* Uncontrolled intercurrent illness.
* Any of the following cardiac abnormalities (only for patients receiving romidepsin):

  1. Congenital long QT syndrome;
  2. corrected QT (QTc) interval ≥ 501 milliseconds;
  3. Patients taking drugs leading to significant QT prolongation (See Appendix 3);
  4. Myocardial infarction within 6 months of cycle 1, day 1. [Subjects with a history of myocardial infarction between 6 and 12 months prior to cycle 1, day 1, who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event, may participate];
  5. Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min);
  6. Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  7. An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥ 2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  8. Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix 5) and/or ejection fraction < 40% by multitargeted acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
  9. A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  10. Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes;
  11. Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
  12. Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers).
* Pregnancy or breast-feeding.
* Active concurrent malignancy (except non-melanoma skin cancer, prostatic intraepithelial neoplasia, or carcinoma in situ of the cervix). Patients whose lymphoma has transformed from a less aggressive histology remain eligible.
* Receipt of solid organ transplant.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis; etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment.
* Central nervous system (CNS) involvement, including lymphomatous meningitis.
* Known active hepatitis A, B or C virus infection.
* Known HIV infection.
* History of primary immunodeficiency.
* Receipt of live, attenuated vaccine within 30 days prior to study entry. Enrolled patients should not receive live vaccine during the study and 30 days after the last dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 year
  The highest dose of study treatment that does not cause unacceptable side effects in patients with R/R PTCL in each study arm

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR will be defined as the sum of complete response rate and partial response rate based on evaluation of best response in each patient.
Duration of Response (DoR) | 1 year
  Time from documentation of tumor response to disease progression
Progression Free Survival (PFS) | 1 year
  Time from study treatment until disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Marchi, M.D., PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No